CLINICAL TRIAL: NCT04530786
Title: Persistence of Influenza Vaccine-induced Antibody in Lung Transplant Patients and Healthy Individuals Beyond the Season
Brief Title: Influenza Vaccine in Lung Transplant Patients - Persistence of Antibodies Beyond the Season
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2004-0240d; A561000 (Other: UW Madison); PHARM/PHARMACY/PHARMACY (Other: UW Madison)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Influenza
Keywords: post-lung transplant; Healthy; immunocompromised
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccine, Post-transplant: Cohort consist of individuals who have received lung transplants Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine
- Vaccine, Healthy Control: Cohort consists of healthy individuals who received the influenza vaccine Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine

INTERVENTIONS:
Drug: Influenza vaccine — influenza vaccine 0.5 ml intramuscularly each season, antigens measured for 3 years following vaccination in:
  * 2004-2005: A/Wyoming H3N2; B/Shanghai
  * 2006-2007: A/New Caledonia H1N1
  * 2007-2008: A/Solomon Islands; A/Wisconsin H3N2; B/Malaysia

SUMMARY:
This a sub-study of a 5-year study designed to investigate how antibody and T cell responses following influenza vaccine compare among lung transplant patients, patients waiting for lung transplantation, and healthy individuals.

This study is designed to investigate influenza vaccine-induced antibodies in lung transplant patients beyond the season of vaccination.

DETAILED DESCRIPTION:
Every year influenza infection causes significant morbidity and mortality in the general population making it a serious public health concern. Among those at highest risk for complications from infection are the immunocompromised. Effective influenza immunization that confers protection throughout the season is critical for lung transplant recipients because in addition to aggressive immunosuppressive therapy, infection directly affects the transplanted organ. Studies of influenza vaccine response rates in lung transplant patients show generally lower antibody concentrations, but acceptable influenza vaccine response rates compared with healthy individuals. However, little is known about the persistence of influenza vaccine-induced antibody concentration in either healthy or immunosuppressed populations.

Influenza antibody concentrations persist at seroprotective levels (defined as antibody concentrations at least 40 hemagglutination units) up to a year post vaccination. However, the investigators could find no information regarding persistence beyond one year.

It is hypothesized that the high rates of persisting influenza vaccine antibody in immunosuppressed lung transplant individuals would match the rates of persisting vaccine-antibody in healthy individuals.

Influenza antibody concentrations against viruses no longer included in the vaccine were measured in serum by hemagglutination inhibition assay (HIA) annually (individual participants followed for 3 years). Samples were collected at 2-4 weeks post-vaccination. Seroprotection was defined as a titer of ≥ 1:40 and was compared between groups over the measured term using Fisher's exact tests.

[This substudy that was originally registered to NCT00205270 and subsequently registered to its own NCT number for the purpose of clarity in linked results]

ELIGIBILITY:
Inclusion Criteria:

* Receiving care Post-lung transplant at University of Wisconsin Hospital
* Healthy adult

Exclusion Criteria:

* Allergy to eggs
* Moderate to severe febrile illness
* Active treatment for acute rejection
* Received season's influenza vaccine prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult or patient receiving care post-lung transplant at the University of Wisconsin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Antibody response to influenza vaccine | season 1 (up to 1 year on study)
  Influenza antibody concentrations against viruses no longer included in the vaccine were measured in serum by hemagglutination inhibition assay (HIA) annually following vaccination of lung transplant participants and healthy controls.
Antibody response to influenza vaccine | season 2 (up to 2 years on study)
  Influenza antibody concentrations against viruses no longer included in the vaccine were measured in serum by hemagglutination inhibition assay (HIA) annually following vaccination of lung transplant participants and healthy controls.
Antibody response to influenza vaccine | season 2 (up to 2.5 years on study)
  Influenza antibody concentrations against viruses no longer included in the vaccine were measured in serum by hemagglutination inhibition assay (HIA) annually following vaccination of lung transplant participants and healthy controls.
Antibody response to influenza vaccine | season 3 (up to 3 years on study)
  Influenza antibody concentrations against viruses no longer included in the vaccine were measured in serum by hemagglutination inhibition assay (HIA) annually following vaccination of lung transplant participants and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Hayney, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Severson JJ, Richards KR, Moran JJ, Hayney MS. Persistence of influenza vaccine-induced antibody in lung transplant patients and healthy individuals beyond the season. Hum Vaccin Immunother. 2012 Dec 1;8(12):1850-3. doi: 10.4161/hv.21735. Epub 2012 Aug 21. PMID 22906937